CLINICAL TRIAL: NCT04090723
Title: Using CBPR to Engage Hazardous Drinking Women in the HIV Prevention and Care Continuum
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00175899; U34AA026220 (NIH)
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: HIV; Alcohol; Harmful Use; Mental Health Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Single Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Computer-delivered brief alcohol intervention (CBI-CC) (Experimental): Participants will be offered only the Computer-delivered brief alcohol intervention with peer navigation from beginning of study to the end.
  Interventions: Behavioral: CBI-CC with peer navigation

INTERVENTIONS:
Behavioral: CBI-CC with peer navigation — Computer delivered brief alcohol intervention enhanced with information of HIV infection, HIV risk, and comorbid mental health disorders

SUMMARY:
Unhealthy alcohol use among women with and at risk for HIV can interrupt critical steps in the HIV prevention and care continuum, is associated with HIV transmission risk behaviors, and contributes to health disparities. Thus it is critical to accurately identify alcohol use and implement alcohol interventions among women with and at risk for HIV to optimize health outcomes. The proposed pilot study will examine the implementation and effects of a computer delivered brief alcohol intervention with peer navigation/Community Health Worker compared to usual care on alcohol use, linkage to health services, and uptake of HIV prevention practices.

DETAILED DESCRIPTION:
Women account for 1 in 4 people living with HIV (PLWH) in the United States, and while African American (AA) women comprise only 14% of the US female population, African American women account for greater than 60% of women living with HIV (WLWH). Unhealthy alcohol use interrupts critical steps in the HIV prevention and care continuum (HPACC) and thus contributes to significant health disparities among at-risk and WLWH. The investigators have developed theory-based, in-person and computer-delivered brief interventions (CBI) for at risk and WLWH with alcohol use, demonstrating drinking reduction. However behavioral and structural barriers to optimal uptake of alcohol interventions and engagement in the HPACC remain, including mental health comorbidity and low knowledge, access, and use of HIV prevention practices such as HIV pre-exposure prophylaxis (PrEP). The goals of this proposal are two-fold: 1) to build on the investigators' current community partnerships to determine how to optimally implement evidence based alcohol treatment for at risk and WLWH in Baltimore, and 2) to determine whether the addition of information, motivational and peer navigator/Community Health Worker support related to comorbid mental health, and HIV prevention practices can enhance CBI and improve alcohol and HPACC outcomes among at risk and WLWH. To achieve these goals the investigators will use a Community Based Participatory Research (CBPR) approach, engaging patient and community stakeholders during all aspects of study development, and community pilot testing. In collaboration with the investigators' Community Advisory Board (CAB), the investigators will: 1) adapt the investigators' current CBI to address gaps in the HIV prevention and care continuum (CBI-CC). The investigators will conduct focus groups with both at risk and WLWH to tailor intervention manuals. 2) The investigators will conduct a pilot study of CBI-CC and peer navigation among 30 at-risk or WLWH with unhealthy alcohol use. The investigators hypothesize that the CBI-CC will result in reduction in drinking and heavy drinking days, increase linkage to substance use, and mental health services and HIV pre exposure prophylaxis (PrEP), and increase use of HIV prevention practices including condoms and PrEP. Through this U34 planning grant the investigators will partner with key stakeholders in the community to build capacity to deliver effective, evidence-based interventions at the nexus of alcohol and HIV for at risk and WLWH with alcohol misuse, and improve engagement in the HIV prevention and care continuum.

ELIGIBILITY:
Inclusion Criteria:

* At risk and Women with HIV ≥18 years
* Alcohol misuse, defined as >7 standard drinks per week or > 3 drinks per occasion in the last three months or AUDIT-C ≥3
* Able to understand English
* Able to read at a 5th grade level.

Additional inclusion criteria for at risk women:

* sex under the influence of alcohol or
* exchanging sex for money or other resources or
* unprotected vaginal or anal sex or illicit drug use in the last 12 months

Exclusion Criteria:

* Pregnant (will be referred immediately to alcohol, mental health, substance use treatment as needed)
* Non-English speaking
* Unable to receive text messages
* Actively psychotic, or otherwise not able to participate in the computer delivered brief intervention.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cis-gender and transgender women will be included
Enrollment: 12 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Intervention Feasibility as assessed by a 4-item scale | 3 months
  Feasibility of the Intervention will be assessed by the Mean/Median score on a 4 item scale that measures the extent to which the new treatment, or an innovation, can be successfully used or carried out within a given agency or setting. Score ranges from 5-20 on the 4 item scale. Higher score means greater feasibility.
Intervention Acceptability as assessed by a 4-item scale | 3 months
  Acceptability of the Intervention will be assessed by the Mean/Median score on a 4 item scale that measures the perception among implementation stakeholders that a given treatment, service, practice, or innovation is agreeable, palatable, or satisfactory. Score ranges from 5-20 on the 4 item scale. Higher score means greater acceptability.

SECONDARY OUTCOMES:
Number of participants linked to services | 3 months
  Linkage to mental health, substance use, HIV pre-exposure prophylaxis or HIV clinical services.
Number of participants with pre-exposure prophylaxis (PrEP) or condom uptake | 3 months
  Uptake of HIV pre-exposure prophylaxis or condoms by participants.
Number of drinking days | At 3 months
  Number of drinking days over past 30 days
Number of heavy drinking days | At 3 months
  Number of heavy drinking days over past 30 days

OTHER OUTCOMES:
Number of condom-less sex episodes | 3 months
  This will be counted to assess sexual risk behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Geetanjali Chander, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No